CLINICAL TRIAL: NCT07094594
Title: Comparing Hartmann's Procedure and Primary Resection With Anastomosis in Hinchey III-IV Diverticulitis: Focus on Ostomy Closure and Long-Term Outcomes
Brief Title: ARES Trial: Approach to Resection and Evaluation in Severe Diverticulitis
Acronym: ARES
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Principal Investigator, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 20251107
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Diverticular Disease of Colon; Colostomy - Stoma; Loop Ileostomies
Keywords: diverticular disease of colon; Hartmann; loop ileostomies
MeSH Terms: conditions — Diverticulosis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hartmann's Procedure Hartmann's Procedure (HP): Hartmann's Procedure (Hartmann's Procedure (HP)): Segmental resection of the sigmoid colon with the creation of an end colostomy.
- Primary Anastomosis and Diverting Loop Ileostomy (PADLI): Primary Anastomosis and Diverting Loop Ileostomy (PADLI): Segmental resection followed by end-to-end anastomosis, protected by a diverting loop ileostomy.

SUMMARY:
This observational study was conducted across five surgical centers in Italy, including both academic and community hospitals, from January 2017 to December 2022. The study aimed to evaluate outcomes in patients with acute perforated sigmoid diverticulitis classified as Hinchey Stage III or IV. All consecutive patients aged 18 years or older who presented with acute perforated sigmoid diverticulitis and underwent emergency colonic resection were included. Patients were excluded if they had Hinchey Stage I or II diverticulitis, postoperative confirmation of malignancy, or underwent laparoscopic surgery. This approach ensured a well-defined patient cohort for consistent and reliable analysis.

DETAILED DESCRIPTION:
This multicenter, prospective observational study evaluated clinical outcomes in adult patients with acute perforated sigmoid diverticulitis classified as Hinchey Stage III or IV, who underwent emergency open colonic resection in five surgical centers in Italy. The study period extended from January 2017 to December 2022 and involved both academic and community hospitals, providing a representative overview of real-world surgical practice.

All consecutive patients aged 18 years or older with a clinical and radiological diagnosis of Hinchey III-IV perforated sigmoid diverticulitis were considered for inclusion. Eligible patients were required to be clinically stable at presentation, enabling them to undergo either primary anastomosis with diverting loop ileostomy or Hartmann's procedure , based on surgeon judgment and intraoperative findings.

Exclusion criteria included:

* Hinchey Stage I or II diverticulitis
* Postoperative confirmation of malignancy as the primary cause of the perforation
* Laparoscopic procedures instead of open resections
* Patients with severe hemodynamic instability, septic shock, or uncontrolled sepsis The primary objective was to compare short- and long-term outcomes between primary anastomosis with diverting loop ileostomy and Hartmann's procedure, including postoperative morbidity and mortality, quality of life, stoma reversal rates, and hospital readmissions. Secondary endpoints included surgical site infections, length of hospital stay, and long-term complications such as parastomal hernia.

This structured design ensured a well-defined and homogeneous study cohort for outcome comparison, allowing for the generation of meaningful real-world evidence on the optimal surgical management of complicated diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Clinical diagnosis of perforated sigmoid diverticulitis (Hinchey Stage III or IV)
* Clinically stable and suitable for undergoing emergency colonic resection
* Eligible to receive either primary anastomosis with diverting loop ileostomy or Hartmann's procedure
* Informed consent provided by the patient or a legal surrogate

Exclusion Criteria:

Hinchey Stage I or II diverticulitis

* Postoperative confirmation of malignancy as the primary cause of perforation
* Laparoscopic surgery instead of open colonic resection
* Unstable patients with severe sepsis, septic shock, or significant hemodynamic compromise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) who presented with acute perforated sigmoid diverticulitis (PSD) classified as Hinchey Stage III or IV and underwent emergency open colonic resection. All participants were clinically stable at the time of surgery and were eligible to receive either primary anastomosis with diverting loop ileostomy (PADLI) or Hartmann's procedure (HP).
  Patients with Hinchey Stage I-II diverticulitis, postoperative confirmation of malignancy, laparoscopic surgery, or hemodynamic instability were excluded to ensure a well-defined and homogeneous study cohort for consistent outcome analysis.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
ostomy closure | 24 mounths
  The primary endpoint was ostomy closure within 24 months, defined as the successful reversal of the stoma. This outcome was chosen as a measure of complete care, reflecting the restoration of bowel continuity and functionality.

SECONDARY OUTCOMES:
Quality of life, assessed using validated tools such as the SF-36 | 24 months
  Quality of life will be evaluated using the Short Form Health Survey (SF-36), a validated questionnaire assessing physical and mental health. The SF-36 score ranges from 0 to 100, with higher scores indicating better quality of life across its domains (physical functioning, role limitations, pain, general health, vitality, social functioning, and mental health).

CONTACTS AND LOCATIONS:
Locations (1):
- Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The decision not to share IPD is based on institutional policies and ethical considerations related to patient confidentiality and data protection. Additionally, no data-sharing infrastructure has been established within the current study protocol, and there are no plans at this time to develop such a framework.